CLINICAL TRIAL: NCT06794385
Title: Comparison of the Effectiveness, Safety, and Satisfaction of Different Methods for Labor Induction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-403/2024-2711-3
Record Dates: First submitted 2025-01-14; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Induction of Labour
Keywords: misoprostol; induction of labour; dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group undergoing labor induction with the dinoprostone vaginal delivery system (Active Comparator): Pregnant women in this group will receive a vaginal delivery system containing 10 mg of dinoprostone for labor induction. The medication will be inserted into the posterior fornix of the vagina, with the active substance being released over a 24-hour period. Maternal and fetal health will be monitored during their stay on the ward. Upon the onset of contractions or any signs of fetal distress, patients will be transferred to the delivery unit. If labor does not commence and the cervix remains unfavorable after 24 hours, a new vaginal delivery system will be inserted for an additional 24 hours. If no progress is observed within 48 hours of induction, a mechanical method for labor induction or cesarean delivery will be employed. After delivery, women will complete a questionnaire to assess their satisfaction with the childbirth experience.
  Interventions: Drug: dinoprostone vaginal delivery system
- Group undergoing labor induction with the low dose peroral misoprostol (Active Comparator): Participants will be induced with a low-dose oral formulation of misoprostol, administered per protocol at 25 mcg every 2 hours until adequate uterine contractions and a favorable cervical condition are achieved. A maximum of 8 doses will be administered on the first day. If labor does not commence and the cervix remains unfavorable, a second induction cycle will be initiated the following day. If no progress occurrs after 48 hours from the induction, participants will undergo cesarean delivery, or alternative mechanical induction method will be used. Following delivery, participants will complete a questionnaire to assess their satisfaction with the childbirth experience.
  Interventions: Drug: low dose peroral misoprostol

INTERVENTIONS:
Drug: dinoprostone vaginal delivery system — Pregnant women in this group will receive a vaginal delivery system containing 10 mg of dinoprostone for labor induction.
  Arms: Group undergoing labor induction with the dinoprostone vaginal delivery system
Drug: low dose peroral misoprostol — Participants will be induced with a low-dose oral formulation of misoprostol, administered per protocol at 25 mcg every 2 hours
  Arms: Group undergoing labor induction with the low dose peroral misoprostol

SUMMARY:
The objective of this interventional study is to compare the effectiveness, safety, and patient satisfaction associated with two commonly used methods of labor induction: low-dose oral misoprostol and the vaginal delivery system with dinoprostone.

The study aims to identify the most suitable induction method for specific subgroups of patients based on parity, body mass index (BMI), age, and cervical ripeness, as well as assess patient preferences for these induction methods.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 37 0/7 and 42 0/7 weeks
* Singleton pregnancy
* Viable fetus in cephalic presentation
* Bishop score ≤ 6
* Maximum parity of three
* Reactive CTG at admission without pathological findings

Exclusion Criteria:

* Age < 18 years
* Gestational age < 37 0/7 weeks
* Active labor
* Spontaneous rupture of membranes
* Non-reassuring CTG findings
* Suspected infection (e.g., fever > 38°C, chorioamnionitis, or unexplained systemic infection)
* Contraindications to vaginal delivery or prostaglandin use
* Previous cesarean delivery or uterine surgery involving entry into the uterine cavity
* Significant fetal abnormalities
* Severe fetal growth restriction with an estimated fetal weight below the 3rd percentile
* Non-Slovenian-speaking participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-01-22 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time from induction to delivery | 1 week from induction
  The time from the insertion of the vaginal delivery system or administration of the oral tablet to the time of delivery

SECONDARY OUTCOMES:
Time from induction to spontaneos vaginal delivery | 1 week from induction
  The time from the insertion of the vaginal delivery system or administration of the oral tablet to the time of spontaneous vaginal delivery
Time from induction to onset of active labour | 1 week from induction
  The investigators will measure the time from the insertion of the vaginal delivery system or administration of the oral tablet to the onset of active labor, defined as the occurrence of strong contractions every 5 minutes.
Use of oxytocin and its dosage | 1 week from induction
  The investigators will compare the need for oxytocin administration and its dosage, measured in international units (IU).
Use of analgesia during labour | 1 week from induction
  The need for epidural analgesia, remifentanil, N₂O, no analgesia.
Type of delivery | 1 week from induction
  Vaginal birth, Caesarean birth, Vacuum extraction
Hyperstimulation with nonreassuring fetal heart rate tracing | 1 week from induction
  Rate of uterine hyperstimulation- exaggerated uterine response consisting of uterine hypertonus, a single uterine contraction lasting two or more minutes or uterine tachysystole with a least 12 contractions in 20 minutes, with a simultaneous nonreassuring fetal heart rate tracing as defined by the 2015 FIGO (The international federation of gynaecology and obstetrics) classification of intrapartum cardiotocography.
Duration of labour | 1 week from induction
  Time from the onset of labor (regular contraction every 5 minutes) to the delivery of the baby
Postpartum hemorrhage above 1000 mL | 1 week from induction
  The investigators will assess whether participants experience blood loss exceeding 1000 mL during delivery and within the first 3 hours postpartum.
Number of participants with third degree tear of perineum during labour | 1 week from induction
  The investigators will observe the occurrence of third-degree perineal tears during labor. A third-degree tear involves injury to the anal sphincter complex, classified as follows: 3a involves less than 50% of the external anal sphincter (EAS) being torn, 3b involves more than 50% of the EAS being torn, and 3c involves tearing of both the EAS and the internal anal sphincter (IAS).
Number of participants with fourth degree tear of perineum during labour | 1 week from induction
  The investigators will observe the occurrence of fourth-degree perineal tears during labor. A fourth-degree tear involves injury to the anal sphincter complex (EAS and IAS) as well as the anorectal mucosa.
Side effects of misoprostol and dinoprostone | 1 week from induction
  The investigators will monitor for the occurrence of the following side effects: nausea, vomiting, high fever, discomfort, diarrhea, and allergic reactions.
Number of newborns wtih 5-minute APGAR score of less than 7 | 1 week from induction
  Infants with a 5-minute APGAR score of less than 7.The Apgar score is a number calculated by scoring the heart rate, respiratory effort, muscle tone, skin color, and reflex irritability of the infant, 5 min after birth. Each of these objective signs can receive 0, 1, or 2 points. The higher is the sum of the points, the better is the condition of the newborn.
  5-minute APGAR score of less than 7.
pH from umbilical artery | 1 week from induction
  A sample will be taken from the umbilical artery after birth for pH analysis.
Number of newborns admitted to intensive care unit | 3 weeks from induction
  Infants which will be admitted to the neonatal intensive unit for whatever reason.
Satisfaction with induction | 1 week from induction
  All participants will complete questionnaires designed to assess whether they experienced any feelings of coercion or undue pressure when consenting to labor induction. These surveys will include four questions specifically focused on labor induction, with responses measured using a Likert scale. The questionnaires will be administered after participants have agreed to proceed with the induction process.
Satisfaction with childbirth | 3 weeks from induction
  The second questionnaire, the validated Childbirth Experience Questionnaire (CEQ2), assesses satisfaction with the labor and delivery process. Participants will complete the CEQ2 within the first three days postpartum while still admitted to the maternity ward. The survey comprises 22 statements specifically addressing aspects of labor induction and the childbirth experience, with responses evaluated using a Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
IPD will be available on request